CLINICAL TRIAL: NCT00892008
Title: Pregabalin (Lyrica) Action In Neuropathic Pain Syndrome (PAINS): A Post Marketing Surveillance Study On Efficacy, Safety And Tolerability Of Pregabalin
Brief Title: A Post Marketing Surveillance Study On Pregabalin (Lyrica) On Efficacy, Safety And Tolerability Of Pregabalin
Acronym: PAINS
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A0081094
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Results first posted 2009-11-18 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2010-01

CONDITIONS: Neuropathic Pain
Keywords: pregabalin; neuropathic pain; safety
MeSH Terms: conditions — Neuralgia | interventions — Pregabalin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Open-Label: This study was open-label with only one treatment group. Pregabalin was prescribed in accordance with usual clinical practice.
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Pregabalin — Pregabalin 75-150 mg BID for at least 2 weeks.
  Other Names: Lyrica

SUMMARY:
This study is being conducted as a regulatory requirement post initial marketing authorization. This is primarily a safety study. This was an open label study and patients were enrolled once the decision to prescribe the medication was made by the Investigator.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years old and above diagnosed with neuropathic pain.

Exclusion Criteria:

* Patients that are pregnant and lactating; and patients with known hypersensitivity to pregabalin or its related components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female, 18 years and above diagnosed with neuropathic pain.
Sampling Method: Non-Probability Sample
Enrollment: 2278 (Actual)
Dates: Start 2006-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081094&StudyName=A%20Post%20Marketing%20Surveillance%20Study%20On%20Pregabalin%20%28Lyrica%29%20On%20Efficacy%2C%20Safety%20And%20Tolerability

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase 4 nationwide post-marketing surveillance study conducted between Sep 2006 and Aug 2008.
Groups:
- Pregabalin: 75-150 milligrams (mg) twice a day (BID) for at least 2 weeks; followed by optional upward dose titration to 600 mg/day at the discretion of the physician/investigator.
Period: Overall Study
Arm/Group | Pregabalin
Started | 2278
Completed | 1713
Not Completed | 565
Not completed — Death | 5
Not completed — Lack of Efficacy | 3
Not completed — Lost to Follow-up | 142
Not completed — Other | 378
Not completed — Adverse Event | 37

BASELINE CHARACTERISTICS:
Arm/Group | Pregabalin
Number analyzed (Participants) | 2278
Age, Customized [Number; unit: participants]
  18-44 years | 582
  45-64 years | 1054
  ≥ 65 years | 451
  unspecified | 191
Sex/Gender, Customized [Number; unit: participants]
  female | 1324
  male | 932
  unspecified | 22

OUTCOME MEASURES:

1. Primary Outcome: Number and Severity of Adverse Events (All Causalities); Baseline to Final Visit (Week 4)
Description: Number and severity of adverse events, including serious adverse events. If the same subject had more than one occurance in the same preferred term event category, only the most severe occurrence was taken.
Time Frame: Baseline through Final Visit (Week 4)
Population: Safety population: all subjects who took at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 2278
participants
  Cardiac Disorders | 1
  palpitations (mild) | 1
  Ear and Labyrinth Disorders | 3
  ear disorder (moderate) | 1
  vertigo (moderate) | 1
  vertigo (severe) | 1
  Gastrointestinal Disorders | 44
  abdominal discomfort (moderate) | 1
  abdominal distension (unspecified) | 1
  abdominal pain (upper) | 1
  constipation (unspecified) | 1
  constipation (mild) | 1
  diarrhoea (mild) | 1
  diarrhoea (moderate) | 1
  dry mouth (mild) | 3
  dry mouth (moderate) | 3
  dyspepsia (mild) | 1
  epigastric discomfort (mild) | 1
  nausea (mild) | 10
  nausea (moderate) | 13
  nausea (severe) | 4
  vomiting (mild) | 8
  vomiting (moderate) | 4
  vomiting (severe) | 1
  General Disorders & Administration Site Conditions | 20
  asthenia (mild) | 2
  asthenia (moderate) | 2
  asthenia (severe) | 1
  fatigue (moderate) | 2
  ill-defined disorder (mild) | 5
  ill-defined disorder (moderate) | 2
  ill-defined disorder (severe) | 1
  irritability (mild) | 2
  irritability (moderate) | 1
  multi-organ failure (unspecified) | 1
  oedema peripheral (unspecified) | 1
  oedema peripheral (moderate) | 1
  pyrexia (mild) | 2
  Hepatobiliary Disorders | 1
  jaundice (moderate) | 1
  Infections and Infestations | 2
  bronchopneumonia (unspecified) | 1
  pneumonia (unspecified) | 1
  Investigations | 1
  weight increased (moderate) | 1
  Metabolism and Nutrition Disorders | 3
  anorexia (moderate) | 1
  hypoglycemia (moderate) | 1
  increased appetite (mild) | 1
  Musculoskeletal and Connective Tissue Disorders | 2
  muscular weakness (mild) | 1
  myalgia (mild) | 1
  Neoplasms Benign, Malignant and Unspecified | 3
  breast cancer stage III (unspecified) | 1
  metastases to central nervous system (unspecified) | 1
  metastatic neoplasm (unspecified) | 1
  Nervous System Disorders | 233
  balance disorder (mild) | 1
  dizziness (unspecified) | 2
  dizziness (mild) | 79
  dizziness (moderate) | 47
  dizziness (severe) | 8
  headache (mild) | 3
  headache (moderate) | 1
  hypersomnia (mild) | 5
  hypersomnia (moderate) | 2
  incoherent (moderate) | 1
  neuralgia (unspecified) | 1
  paraesthesia (mild) | 1
  sedation (moderate) | 3
  sedation (severe) | 2
  somnolence (unspecified) | 3
  somnolence (mild) | 62
  somnolence (moderate) | 24
  somnolence (severe) | 4
  syncope (moderate) | 1
  syncope (severe) | 1
  tremor (moderate) | 1
  Psychiatric Disorders | 3
  abnormal dreams (moderate) | 1
  confusional state (mild) | 1
  insomnia (severe) | 1
  Reproductive and Breast Disorders | 1
  ejaculation disorder (unspecified) | 1
  Respiratory, Thoracic and Mediastinal Disorders | 3
  dyspnoea (severe) | 1
  dyspnoea exertional (mild) | 1
  snoring (severe) | 1
  Skin and Subcutaneous Tissue Disorders | 1
  rash generalized (severe) | 1
  Vascular Disorders | 3
  hypertension (unspecified) | 1
  hypotension (moderate) | 1
  pallor (mild) | 1

2. Secondary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score
Description: Change from Baseline in 10 cm VAS pain score; 10-point pain intensity ordinal rating system: 0 = no pain, 1-3 = mild pain, 4-6 = moderate pain, 7-9 = severe pain, 10 = worst possible pain. Change = scores at second visit and final visit minus score at Baseline.
Time Frame: Baseline, Second Visit (Week ≥ 2), Final Visit (Week 4)
Population: Intent to treat (ITT) population: a subset of the safety population who underwent Baseline assessment, received study drug for at least 2 weeks, and had at least 1 follow-up visit. N = number of subjects with a Visual Analog Scale (VAS) pain score at Baseline Visit.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 1558
scores on scale
  Second Visit (n=1472) | 3.5 (1.7)
  Final Visit (n=1126) | 5.1 (1.8)

3. Secondary Outcome: VAS Pain Score at Baseline (BL) and Second Visit
Description: VAS Pain Score: 10 cm (10-point) pain intensity ordinal rating system: 0 = no pain, 1-3 = mild pain, 4-6 = moderate pain, 7-9 = severe pain, 10 = worst possible pain. Shift table shows the number of subjects with each pain intensity rating at the Second Visit by the number of subjects with each pain intensity rating at Baseline. Abbreviations: mod = moderate, sev = severe, wrst = worst, poss = possible, pn = pain, vst = visit .
Time Frame: Baseline, Second Visit (Week ≥ 2)
Population: Intent to treat (ITT) population: a subset of the safety population who underwent Baseline assessment, received study drug for at least 2 weeks, and had at least 1 follow-up visit. N=number of subjects in ITT population.
Measure: Number; unit: participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 1603
participants
  BL: Mild Pain (n=25); 2nd Visit: Mild Pain | 22
  BL: Mild Pain (n= 25); 2nd Visit: Moderate Pain | 0
  BL: Mild Pain (n= 25); 2nd Visit: Severe Pain | 0
  BL:Mild Pain (n= 25); 2nd Visit: Worst Poss. Pain | 0
  BL: Mild Pain (n= 25); 2nd Visit: Missing | 3
  BL: Moderate Pain (n=450); 2nd Visit: Mild Pain | 300
  BL: Moderate Pain (n=450): 2nd Visit: Mod Pain | 115
  BL: Moderate Pain (n=450); 2nd Visit: Severe Pain | 2
  BL: Mod Pain (n=450); 2nd Visit: Worst Poss. Pain | 0
  BL: Moderate Pain (n=450); 2nd Visit: Missing | 33
  BL: Severe Pain (n=985); 2nd Visit: Mild Pain | 348
  BL: Severe Pain (n=985); 2nd Visit: Moderate Pain | 533
  BL: Severe Pain (n=985) ; 2nd Visit: Severe Pain | 59
  BL: Sev Pain (n=985); 2nd Visit: Worst Poss. pain | 0
  BL: Severe Pain (n=985); 2nd Visit: Missing | 45
  BL: Worst Poss. Pain (n=98) ; 2nd Visit: Mild Pain | 18
  BL: Worst Poss. Pain (n=98); 2nd Visit: Mod Pain | 49
  BL: Worst Poss. Pain (n=98); 2nd Visit: Sev Pain | 25
  BL:Wrst Poss Pain (n=98); 2nd Visit: Wrst Poss. Pn | 1
  BL: Worst Poss. Pain (n=98) ; 2nd Visit: Missing | 5
  BL: Missing (n=45); 2nd Visit: Mild Pain | 3
  BL: Missing (n=45) ; 2nd Visit: Moderate Pain | 1
  BL: Missing (n=45) ; 2nd Visit: Severe Pain | 3
  BL: Missing (n=45) ; 2nd Visit: Worst Poss. Pain | 0
  BL: Missing (n=45); 2nd Visit: Missing | 38

4. Secondary Outcome: VAS Pain Score at Baseline and Final Visit
Description: VAS Pain Score 10 cm (10-point) pain intensity ordinal rating system: 0 = no pain, 1-3 = mild pain, 4-6 = moderate pain, 7-9 = severe pain, 10 = worst possible pain. Shift table shows the number of subjects with each pain intensity rating at the Final Visit by the number of subjects with each pain intensity rating at Baseline. Abbreviations: mod = moderate, sev = severe, wrst = worst, poss = possible, pn = pain, vst = visit.
Time Frame: Baseline, Final Visit (Week 4)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 1603
participants
  BL: Mild Pain (n=25); Final Visit: Mild Pain | 12
  BL: Mild Pain (n=25); Final Visit: Moderate Pain | 0
  BL: Mild Pain (n=25); Final Visit: Severe Pain | 0
  BL: Mild Pain (n=25); Final Visit: Missing | 13
  BL: Moderate Pain (n=450); Final Visit: Mild Pain | 272
  BL: Moderate Pain (n=450); Final Visit: Mod. Pain | 19
  BL: Moderate Pain (n=450); Final Visit: Sev. Pain | 1
  BL: Moderate Pain (n=450); Final Visit: Missing | 158
  BL: Severe Pain (n=985); Final Visit: Mild Pain | 602
  BL: Severe Pain (n=985); Final Visit: Mod. Pain | 134
  BL: Severe Pain (n=985); Final Visit: Severe Pain | 6
  BL: Severe Pain (n=985); Final Visit: Missing | 243
  BL: Worst Poss. Pain (n=98); Final Vst: Mild Pain | 54
  BL: Worst Poss. Pain (n=98); Final Vst: Mod Pain | 25
  BL: Worst Poss. Pain (n=98); Final Visit: Sev Pain | 1
  BL: Worst Poss. Pain (n=98); Final Visit: Missing | 18
  BL: Missing (n=45); Final Visit: Mild Pain | 4
  BL: Missing (n=45); Final Visit: Moderate Pain | 1
  BL: Missing (n=45); Final Visit: Severe Pain | 1
  BL: Missing (n=45); Final Visit: Missing | 39

5. Secondary Outcome: Physician's Clinical Global Impression (CGI) of Treatment Satisfaction at the Second and Final Visits
Description: Physician's Clinical Global Impression of treatment satisfaction. Treatment satisfaction item of the CGI has a scale of five discrete score points: excellent, very good, good, fair and poor. Shift table shows the number of subjects with each score point rating at the Final Visit by the number of subjects with each score point rating at the Second Visit.
Time Frame: Second Visit (Week ≥ 2), Final Visit (Week 4)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 1603
participants
  2nd Visit: Excellent (n=272); Final Vst: Excellent | 209
  2nd Visit: Excellent (n=272); Final Vst: Very Good | 6
  2nd Visit: Excellent (n=272); Final Visit: Good | 2
  2nd Visit: Excellent (n=272); Final Visit: Fair | 0
  2nd Visit: Excellent (n=272); Final Visit: Poor | 0
  2nd Visit: Excellent (n=272); Final Visit: Missing | 55
  2nd Visit: Very Good (n=803); Final Vst: Excellent | 307
  2nd Visit: Very Good (n=803); Final Vst: Very Good | 421
  2nd Visit: Very Good (n=803); Final Visit: Good | 10
  2nd Visit: Very Good (n=803); Final Visit: Fair | 0
  2nd Visit: Very Good (n=803); Final Visit: Poor | 0
  2nd Visit: Very Good (n=803); Final Visit: Missing | 65
  2nd Visit: Good (n=438); Final Visit: Excellent | 27
  2nd Visit: Good (n=438); Final Visit: Very Good | 267
  2nd Visit: Good (n=438); Final Visit: Good | 119
  2nd Visit: Good (n=438); Final Visit: Fair | 4
  2nd Visit: Good (n=438); Final Visit: Poor | 0
  2nd Visit: Good (n=438); Final Visit: Missing | 21
  2nd Visit: Fair (n=71); Final Visit: Excellent | 7
  2nd Visit: Fair (n=71); Final Visit: Very Good | 22
  2nd Visit: Fair (n=71); Final Visit: Good | 30
  2nd Visit: Fair (n=71); Final Visit: Fair | 3
  2nd Visit: Fair (n=71); Final Visit: Poor | 1
  2nd Visit: Fair (n=71); Final Visit: Missing | 8
  2nd Visit: Poor (n=7); Final Visit: Excellent | 0
  2nd Visit: Poor (n=7); Final Visit: Very Good | 1
  2nd Visit: Poor (n=7); Final Visit: Good | 2
  2nd Visit: Poor (n=7); Final Visit: Fair | 1
  2nd Visit: Poor (n=7); Final Visit: Poor | 1
  2nd Visit: Poor (n=7); Final Visit: Missing | 2
  2nd Visit: Missing (n=12); Final Visit: Excellent | 0
  2nd Visit: Missing (n=12); Final Visit: Very Good | 0
  2nd Visit: Missing (n=12); Final Visit: Good | 0
  2nd Visit: Missing (n=12); Final Visit: Fair | 0
  2nd Visit: Missing (n=12); Final Visit: Poor | 0
  2nd Visit: Missing (n=12); Final Visit: Missing | 12

6. Secondary Outcome: Patient's Clinical Global Impression (CGI) of Treatment Satisfaction at the Second and Final Visits
Description: Patient's Clinical Global Impression of treatment satisfaction. Treatment satisfaction item of CGI has a scale of five discrete points: excellent, very good, good, fair and poor. Shift table shows the number of subjects with each score point rating at the Final Visit by the number of subjects with each score point rating at the Second Visit.
Time Frame: Second Visit (Week ≥ 2), Final Visit (Week 4)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 1603
participants
  2nd Visit: Excellent (n=260); Final Vst: Excell | 201
  2nd Visit: Excell (n=260) ; Final Vst:Very Good | 11
  2nd Visit: Excellent (n=260); Final Visit: Good | 1
  2nd Visit: Excellent (n=260) ; Final Visit: Fair | 0
  2nd Visit: Excellent (n=260) ; Final Visit: Poor | 0
  2nd Visit: Excellent (n=260); Final Visit: Missing | 47
  2nd Visit: Very Good (n=778); Final Visit: Excell | 297
  2nd Visit: Very Good (n=778); Final Vst: Very Good | 394
  2nd Visit: Very Good (n=778); Final Visit: Good | 13
  2nd Visit: Very Good (n=778); Final Visit: Fair | 1
  2nd Visit: Very Good (n=778); Final Visit: Poor | 0
  2nd Visit: Very Good (n=778); Final Visit: Missing | 73
  2nd Visit: Good (n=454); Final Visit: Excellent | 35
  2nd Visit: Good (n=454); Final Visit: Very Good | 263
  2nd Visit: Good (n=454); Final Visit: Good | 130
  2nd Visit: Good (n=454); Final Visit: Fair | 4
  2nd Visit: Good (n=454); Final Visit: Poor | 0
  2nd Visit: Good (n=454); Final Visit: Missing | 22
  2nd Visit: Fair (n=81); Final Visit: Excellent | 9
  2nd Visit: Fair (n=81); Final Visit: Very Good | 23
  2nd Visit: Fair (n=81); Final Visit:: Good | 31
  2nd Visit: Fair (n=81); Final Visit: Fair | 9
  2nd Visit: Fair (n=81); Final Visit: Poor | 1
  2nd Visit: Fair (n=81); Final Visit: Missing | 8
  2nd Visit: Poor (n=12); Final Visit: Excellent | 1
  2nd Visit: Poor (n=12); Final Visit: Very Good | 2
  2nd Visit: Poor (n=12); Final Visit: Good | 2
  2nd Visit: Poor (n=12); Final Visit: Fair | 2
  2nd Visit::Poor (n=12); Final Visit: Poor | 2
  2nd Visit: Poor (n=12); Final Visit: Missing | 3
  2nd Visit: Missing (n=18); Final Visit: Excellent | 0
  2nd Visit: Missing (n=18); Final Visit: Very Good | 2
  2nd Visit: Missing (n=18); Final Visit: Good | 0
  2nd Visit: Missing (n=18); Final Visit: Fair | 1
  2nd Visit: Missing (n=18); Final Visit: Poor | 0
  2nd Visit: Missing (n=18); Final Visit: Missing | 15

7. Secondary Outcome: Physician's Clinical Global Impression (CGI) of Efficacy at Second and Final Visit
Description: Physician's Clinical Global Impression of efficacy. Efficacy item of the CGI has a scale of five discrete points: excellent, very good, good, fair and poor. Shift table shows the number of subjects with each score point rating at the Final Visit by the number of subjects with each score point rating at the Second Visit.
Time Frame: Second Visit (Week ≥ 2), Final Visit (Week 4)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 1603
participants
  2nd Visit: Excellent (n=279); Final Visit: Excell | 217
  2nd Visit: Excellent (n=279); Final Vst: Very Good | 8
  2nd Visit: Excellent (n=279); Final Visit: Good | 1
  2nd Visit: Excellent (n=279); Final Visit: Fair | 0
  2nd Visit: Excellent (n=279); Final Visit: Poor | 0
  2nd Visit: Excellent (n=279); Final Visit: Missing | 53
  2nd Visit: Very Good (n=813); Final Visit: Excell | 298
  2nd Visit: Very Good (n=813); Final Vst: Very Good | 437
  2nd Visit: Very Good (n=813); Final Visit: Good | 10
  2nd Visit: Very Good (n=813); Final Visit: Fair | 0
  2nd Visit: Very Good (n=813); Final Visit: Poor | 0
  2nd Visit: Very Good (n=813); Final Visit: Missing | 68
  2nd Visit: Good (n=418); Final Visit: Excellent | 19
  2nd Visit: Good (n=418); Final Visit: Very Good | 258
  2nd Visit: Good (n=418); Final Visit: Good | 115
  2nd Visit: Good (n=418); Final Visit: Fair | 5
  2nd Visit: Good (n=418); Final Visit: Poor | 0
  2nd Visit: Good (n=418); Final Visit: Missing | 21
  2nd Visit: Fair (n=66); Final Visit: Excellent | 4
  2nd Visit: Fair (n=66); Final Visit: Very Good | 20
  2nd Visit: Fair (n=66); Final Visit: Good | 28
  2nd Visit: Fair (n=66); Final Visit: Fair | 5
  2nd Visit: Fair (n=66); Final Visit: Poor | 2
  2nd Visit: Fair (n=66); Final Visit: Missing | 7
  2nd Visit: Poor (n=7); Final Visit: Excellent | 0
  2nd Visit: Poor (n=7); Final Visit: Very Good | 2
  2nd Visit: Poor (n=7); Final Visit: Good | 2
  2nd Visit: Poor (n=7); Final Visit: Fair | 0
  2nd Visit: Poor (n=7); Final Visit: Poor | 1
  2nd Visit: Poor (n=7); Final Visit: Missing | 2
  2nd Visit: Missing (n=20); Final Visit: Excellent | 0
  2nd Visit: Missing (n=20); Final Visit: Very Good | 1
  2nd Visit: Missing (n=20); Final Visit: Good | 0
  2nd Visit: Missing (n=20); Final Visit: Fair | 0
  2nd Visit: Missing (n=20); Final Visit: Poor | 0
  2nd Visit: Missing (n=20); Final Visit: Missing | 19

8. Secondary Outcome: Patient's Clinical Global Impression (CGI) of Efficacy at Second and Final Visit
Description: Patient's Clinical Global Impression of efficacy. Efficacy item of CGI has a scale of five discrete points: excellent, very good, good, fair and poor. Shift table shows the number of subjects with each score point rating at the Final Visit by the number of subjects with each score point rating at the Second Visit.
Time Frame: Second Visit (Week ≥ 2), Final Visit (Week 4)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 1603
participants
  2nd Visit: Excellent (n=264); Final Visit: Excell | 206
  2nd Visit: Excellent (n=264); Final Vst: Very Good | 8
  2nd Visit: Excellent (n=264); Final Visit: Good | 0
  2nd Visit: Excellent (n=264); Final Visit: Fair | 0
  2nd Visit: Excellent (n=264); Final Visit: Poor | 0
  2nd Visit: Excellent (n=264); Final Visit: Missing | 50
  2nd Visit: Very Good (n=775); Final Visit: Excell | 286
  2nd Visit: Very Good (n=775); Final Vst: Very Good | 405
  2nd Visit: Very Good (n=775); Final Visit: Good | 12
  2nd Visit: Very Good (n=775); Final Visit: Fair | 1
  2nd Visit: Very Good (n=775); Final Visit: Poor | 0
  2nd Visit: Very Good (n=775); Final Visit: Missing | 71
  2nd Visit: Good (n=450); Final Visit: Excellent | 34
  2nd Visit: Good (n=450): Final Visit: Very Good | 266
  2nd Visit: Good (n=450); Final Visit: Good | 127
  2nd Visit: Good (n=450); Final Visit: Fair | 1
  2nd Visit: Good (n=450); Final Visit: Poor | 0
  2nd Visit: Good (n=450); Final Visit: Missing | 22
  2nd Visit: Fair (n=75); Final Visit: Excellent | 6
  2nd Visit: Fair (n=75); Final Visit: Very Good | 21
  2nd Visit: Fair (n=75); Final Visit: Good | 32
  2nd Visit: Fair (n=75); Final Visit: Fair | 10
  2nd Visit: Fair (n=75); Final Visit: Poor | 0
  2nd Visit: Fair (n=75); Final Visit: Missing | 6
  2nd Visit: Poor (n=12); Final Visit: Excellent | 1
  2nd Visit :Poor (n=12); Final Visit: Very Good | 2
  2nd Visit: Poor (n=12); Final Visit: Good | 2
  2nd Visit: Poor (n=12); Final Visit: Fair | 0
  2nd Visit: Poor (n=12); Final Visit: Poor | 3
  2nd Visit: Poor (n=12); Final Visit: Missing | 4
  2nd Visit: Missing (n=27); Final Visit: Excellent | 0
  2nd Visit: Missing (n=27); Final Visit: Very Good | 3
  2nd Visit: Missing (n=27); Final Visit: Good | 0
  2nd Visit: Missing (n=27); Final Visit: Fair | 1
  2nd Visit: Missing (n=27); Final Visit: Poor | 0
  2nd Visit: Missing (n=27); Final Visit: Missing | 23

9. Secondary Outcome: Physician's Clinical Global Impression (CGI) on Tolerability at Second and Final Viist
Description: Physician's Clinical Global Impression of tolerability. Tolerability item of CGI has a scale of five discrete points: excellent, very good, good, fair and poor. Shift table shows the number of subjects with each score point rating at the Final Visit by the number of subjects with each score point rating at the Second Visit.
Time Frame: Second Visit (Week ≥ 2), Final Visit (Week 4)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 1603
participants
  2nd Visit: Excellent (n=309); Final Visit: Excell | 237
  2nd Visit: Excellent (n=309); Final Vst: Very Good | 12
  2nd Visit: Excellent (n=309); Final Visit: Good | 0
  2nd Visit: Excellent (n=309); Final Visit: Fair | 0
  2nd Visit: Excellent (n=309); Final Visit: Poor | 0
  2nd Visit: Excellent (n=309); Final Visit: Missing | 60
  2nd Visit: Very Good (n=764); Final Visit: Excell | 255
  2nd Visit: Very Good (n=764); Final Vst:Very Good | 431
  2nd Visit: Very Good (n=764); Final Visit: Good | 9
  2nd Visit: Very Good (n=764); Final Visit: Fair | 1
  2nd Visit: Very Good (n=764); Final Visit: Poor | 1
  2nd Visit: Very Good (n=764); Final Visit: Missing | 67
  2nd Visit: Good (n=436); Final Visit: Excellent | 24
  2nd Visit: Good (n=436); Final Visit: Very Good | 254
  2nd Visit: Good (n=436); Final Visit: Good | 135
  2nd Visit: Good (n=436); Final Visit: Fair | 1
  2nd Visit: Good (n=436); Final Visit: Poor | 1
  2nd Visit: Good (n=436); Final Visit: Missing | 21
  2nd Visit: Fair (n=67); Final Visit: Excellent | 6
  2nd Visit: Fair (n=67); Final Visit: Very Good | 19
  2nd Visit: Fair (n=67); Final Visit: Good | 30
  2nd Visit: Fair (n=67); Final Visit: Fair | 5
  2nd Visit: Fair (n=67); Final Visit: Poor | 1
  2nd Visit: Fair (n=67); Final Visit: Missing | 6
  2nd Visit: Poor (n=6); Final Visit: Excellent | 1
  2nd Visit: Poor (n=6); Final Visit: Very Good | 0
  2nd Visit: Poor (n=6); Final Visit: Good | 1
  2nd Visit: Poor (n=6); Final Visit: Fair | 0
  2nd Visit: Poor (n=6); Final Visit: Poor | 3
  2nd Visit: Poor (n=6); Final Visit: Missing | 1
  2nd Visit: Missing (n=21); Final Visit: Excellent | 1
  2nd Visit: Missing (n=21); Final Visit: Very Good | 2
  2nd Visit: Missing (n=21); Final Visit: Good | 0
  2nd Visit: Missing (n=21); Final Visit: Fair | 0
  2nd Visit: Missing (n=21); Final Visit: Poor | 0
  2nd Visit: Missing (n=21); Final Visit: Missing | 18

10. Secondary Outcome: Patient's Clinical Global Impression (CGI) of Tolerability at Second and Final Visit
Description: Patient's Clinical Global Impression of tolerability. The tolerability item of CGI has a scale of five discrete points: excellent, very good, good, fair and poor. Shift table shows the number of subjects with each score point rating at the Final Visit by the number of subjects with each score point rating at the Second Visit. Abbreviation: vst = visit.
Time Frame: Second Visit (Week ≥ 2), Final Visit (Week 4)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 1603
participants
  2nd Visit: Excellent (n=278); Final Visit: Excell | 213
  2nd Visit: Excellent (n=278); Final Vst: Very Good | 14
  2nd Visit: Excellent (n=278); Final Visit: Good | 0
  2nd Visit: Excellent (n=278); Final Visit: Fair | 0
  2nd Visit: Excellent (n=278); Final Visit: Poor | 0
  2nd Visit: Excellent (n=278); Final Visit: Missing | 51
  2nd Visit: Very Good (n=750); Final Visit: Excell | 257
  2nd Visit: Very Good (n=750); Final Vst: Very Good | 415
  2nd Visit: Very Good (n=750); Final Visit: Good | 13
  2nd Visit: Very Good (n=750); Final Visit: Fair | 1
  2nd Visit: Very Good (n=750); Final Visit: Poor | 0
  2nd Visit: Very Good (n=750); Final Visit: Missing | 64
  2nd Visit: Good (n=465); Final Visit: Excellent | 27
  2nd Visit: Good (n=465); Final Visit: Very Good | 255
  2nd Visit: Good (n=465); Final Visit: Good | 151
  2nd Visit: Good (n=465); Final Visit: Fair | 4
  2nd Visit: Good (n=465); Final Visit: Poor | 2
  2nd Visit: Good (n=465); Final Visit: Missing | 26
  2nd Visit: Fair (n=71); Final Visit: Excellent | 8
  2nd Visit: Fair (n=71); Final Visit: Very Good | 18
  2nd Visit: Fair (n=71); Final Visit: Good | 31
  2nd Visit: Fair (n=71); Final Visit: Fair | 7
  2nd Visit: Fair (n=71); Final Visit: Poor | 1
  2nd Visit: Fair (n=71); Final Visit: Missing | 6
  2nd Visit: Poor (n=11); Final Visit: Excellent | 1
  2nd Visit: Poor (n=11); Final Visit: Very Good | 2
  2nd Visit: Poor (n=11); Final Visit: Good | 1
  2nd Visit: Poor (n=11); Final Visit: Fair | 0
  2nd Visit: Poor (n=11); Final Visit: Poor | 3
  2nd Visit: Poor (n=11); Final Visit: Missing | 4
  2nd Visit: Missing (n=28); Final Visit: Excellent | 1
  2nd Visit: Missing (n=28); Final Visit: Very Good | 2
  2nd Visit: Missing (n=28); Final Visit: Good | 0
  2nd Visit: Missing (n=28); Final Visit: Fair | 1
  2nd Visit: Missing (n=28); Final Visit: Poor | 0
  2nd Visit: Missing (n=28); Final Visit: Missing | 24

11. Primary Outcome: Discontinuations Due to Adverse Events
Description: Discontinuations due to adverse events by MedDRA system organ class and preferred term.
Time Frame: Baseline, Second Visit (Week ≥ 2), Final Visit (Week 4)
Population: Safety population: all subjects who took at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 2278
participants
  Cardiac Disorders: palpitations | 1
  Ear and Labyrinth Disorders: vertigo | 1
  Gastrointestinal Disorders: nausea | 5
  Gastrointestinal Disorders: vomiting | 3
  General/ Administrative Site Conditions: asthenia | 2
  Nervous System Disorders: somnolence | 26
  Resp., Thoracic & Mediastinal Disorders: snoring | 1
  Vascular Disorders: hypertension | 1

ADVERSE EVENTS:
Time Frame: Adverse events: Baseline through end of study (>= Week 4); serious adverse events: Baseline through and including 28 calendar days after the last administration of study medication (last administration was up to Week 4).
Arm/Group | Pregabalin
Serious Adverse Events (participants affected / at risk) | 7/2278
Other Adverse Events (participants affected / at risk) | 345/2278
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=2278)
Asthenia (General disorders) | 1
Multi-organ failure (General disorders) | 1
Bronchopneumonia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Breast cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Sedation (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=2278)
Palpitations (Cardiac disorders) | 1
Ear disorder (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 6
Dyspepsia (Gastrointestinal disorders) | 1
Epigastric discomfort (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 27
Vomiting (Gastrointestinal disorders) | 13
Asthenia (General disorders) | 4
Fatigue (General disorders) | 2
Ill-defined disorder (General disorders) | 8
Irritability (General disorders) | 3
Oedema peripheral (General disorders) | 2
Pyrexia (General disorders) | 2
Jaundice (Hepatobiliary disorders) | 1
Weight increased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Increased appetite (Metabolism and nutrition disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Balance disorder (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 135
Headache (Nervous system disorders) | 4
Hypersomnia (Nervous system disorders) | 7
Incoherent (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Sedation (Nervous system disorders) | 4
Somnolence (Nervous system disorders) | 92
Syncope (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 1
Abnormal dreams (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Ejaculation disorder (Reproductive system and breast disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Snoring (Respiratory, thoracic and mediastinal disorders) | 1
Rash generalized (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Pallor (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.